CLINICAL TRIAL: NCT05305586
Title: Comparison of Bulk-fill Flowable and Packable Composite in Splinting of Luxation Injuries: A Randomised Control Trial
Brief Title: Comparison of Two Types of Splints to Treat Dental Luxation Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Arshad Hasan, Head of Department, Operative Dentistry, Dow Dental College, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUHS/BASR/2019/472
Record Dates: First submitted 2022-03-04; First posted 2022-03-31 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Dental Trauma; Splints
Keywords: Dental trauma; Splints; bulkfill composite; packable composite

STUDY DESIGN:
Intervention Model Description: The study model was a randomised control trial. The included patients were randomly allocated to either group by a lottery method.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants were unaware of the group allocation. In addition, the outcome assessments were performed by a blinded investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Packable Composite (Active Comparator): Packable composite material was selected for splinting of luxated teeth
  Interventions: Device: Splint retained by Packable Composite
- Bulkfill composite (Active Comparator): Bulkfill composite material was selected for the splinting of luxated teeth
  Interventions: Device: Splint retained by Bulk-fill flowable

INTERVENTIONS:
Device: Splint retained by Bulk-fill flowable — Luxated teeth were splinted with bulk-fill flowable composite
  Arms: Bulkfill composite
Device: Splint retained by Packable Composite — Luxated teeth were splinted with packable composite
  Arms: Packable Composite

SUMMARY:
The objectives of this randomized clinical trial (RCT) were:

1. To compare the efficiency of splinting by two composite materials in terms of retention of material
2. To compare adhesive point dimension between the two groups
3. To compare time taken to place and remove the splint
4. To assess the efficacy of bulkfill flowable in reducing mobility of luxated teeth.

DETAILED DESCRIPTION:
A Randomized control trial of 6 month period was done. Patients with luxation injuries aged between 16- 50 years were asked to participate in the study after taking informed consent. They were then assigned to either group (Group 1: Packable Composite (PC), Group 2: Bulkfill Flowable) by lottery method. Periotest was used to check the mobility of teeth before the placement of splint. Splinting was performed with composite material according to group allocation. Time taken to place the splint was recorded. Frontal view images of splinted teeth were taken with DSLR and transferred to Adobe Photoshop Version 22.4.1 for windows to measure surface area of the restorative material in percentage to total tooth surface area. Post-operative instructions were given. After 2 weeks, Periotest readings were recorded, immediately after removal of splint. On both visits 3 readings per tooth were recorded. Time taken to remove the splint was also recorded. Additionally, the retention of splint was also observed.

STATISTICAL ANALYSIS:

SPSS version 26 for windows was used, the mean time taken to apply and remove the material and mobility before and after removal of splint was compared using the independent samples T test. Mann-Whitney test compared the percentage area of the material occupied. Fisher's Eaxct test evaluated the retention of splint material. Level of significance was kept at p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition patients aged between 16-50 years
* Either gender
* Lateral and extrusive luxation injuries

Exclusion Criteria:

* Patients with following conditions were excluded
* Intrusion injuries
* Root fracture
* Dentoalveolar fracture.
* Patients with systemic diseases.
* Patients with periodontitis
* Para-Functional habits
* Non-consenting patients

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Retention of splint | 2 weeks
  Retention will be measured as follows:
  Fully bonded: No exposure of wire on composite material and wire remained bonded to tooth.
  Partially debonded: Specs of composite remained on wire and wire remained bonded to tooth.
  Unbonded: wire is exposed to oral cavity with no composite on it and wire is detatched from tooth and freely movable.
  The outcome will be measured as percentage of cases reporting with condition of interest in each group.
Adhesive point dimension | 2 weeks
  Percentage of area occupied by the material in comparison to the tooth will be noted as adhesive point dimension.
  The outcome will be measured as percentage occupied by the splinting material of total tooth area as it is visible from the front. In our case the wire splint is retained by either Bulkfill composite or Packable composite. Therefore, the percentage of area occupied by the splinting material is the outcome of interest.
Tooth mobility | 2 weeks
  'Movement of tooth in its socket resulting from an applied force, usually measured on an increasing scale of 1-3, or measured by the amount of horizontal and/or vertical mobility in millimeters'
  The values of Periotest in assessment of tooth mobility is based on the scale given as:
  Grade 0: -0.8- +09 Grade I: +10- +19 Grade II: +20- +29 Grade III: +30- +50
  The outcome will be measured as percentage of patients presenting with grade of tooth mobility before applying the splint and after removal of splint
Time consumed to apply and remove the splint | 2 weeks
  Application time: Amount of time taken in minutes from the beginning of splinting that is starting from applying the etchant till the last block of composite is cured.
  Removal time: The amount of time taken in minutes to remove the splinting material
  The outcome will be measured as amount time taken in mm:ss i.e. minute:second to apply and remove the splint in either group.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Hasan, BDS, FCPS, Study Director — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bratteberg M, Thelen DS, Klock KS, Bardsen A. Traumatic dental injuries-Prevalence and severity among 16-year-old pupils in western Norway. Dent Traumatol. 2018 Jun;34(3):144-150. doi: 10.1111/edt.12399. PMID 29569840
- [Background] Zhu Y, Chen H, Cen L, Wang J. Influence of abutment tooth position and adhesive point dimension on the rigidity of a dental trauma wire-composite splint. Dent Traumatol. 2016 Jun;32(3):225-30. doi: 10.1111/edt.12241. Epub 2015 Oct 28. PMID 26511774
- [Background] Da Silva AC, Passeri LA, Mazzonetto R, De Moraes M, Moreira RW. Incidence of dental trauma associated with facial trauma in Brazil: a 1-year evaluation. Dent Traumatol. 2004 Feb;20(1):6-11. doi: 10.1111/j.1600-4469.2004.00212.x. PMID 14998409
- [Background] Bourguignon C, Cohenca N, Lauridsen E, Flores MT, O'Connell AC, Day PF, Tsilingaridis G, Abbott PV, Fouad AF, Hicks L, Andreasen JO, Cehreli ZC, Harlamb S, Kahler B, Oginni A, Semper M, Levin L. International Association of Dental Traumatology guidelines for the management of traumatic dental injuries: 1. Fractures and luxations. Dent Traumatol. 2020 Aug;36(4):314-330. doi: 10.1111/edt.12578. Epub 2020 Jul 17. PMID 32475015
- [Background] Berthold C, Auer FJ, Potapov S, Petschelt A. Rigidity evaluation of quartz-fiber splints compared with wire-composite splints. Dent Traumatol. 2012 Feb;28(1):65-74. doi: 10.1111/j.1600-9657.2011.01031.x. Epub 2011 Jul 26. PMID 21790986
- [Background] Kaste LM, Gift HC, Bhat M, Swango PA. Prevalence of incisor trauma in persons 6-50 years of age: United States, 1988-1991. J Dent Res. 1996 Feb;75 Spec No:696-705. doi: 10.1177/002203459607502S09. PMID 8594093
- [Background] Khan NA, Qazi HS, Maxood A, Khan AM, Abbas I. Traumatic injuries of the permanent maxillory incisors at Dental Department, Pakistan Institute of Medical Sciences Islamabad: a retrospective study. J Ayub Med Coll Abbottabad. 2008 Jul-Sep;20(3):84-7. PMID 19610526
- [Background] Petti S, Andreasen JO, Glendor U, Andersson L. The fifth most prevalent disease is being neglected by public health organisations. Lancet Glob Health. 2018 Oct;6(10):e1070-e1071. doi: 10.1016/S2214-109X(18)30380-2. No abstract available. PMID 30223983
- [Background] Piovesan C, Abella C, Ardenghi TM. Child oral health-related quality of life and socioeconomic factors associated with traumatic dental injuries in schoolchildren. Oral Health Prev Dent. 2011;9(4):405-11. PMID 22238740
- [Background] Feliciano KM, de Franca Caldas A Jr. A systematic review of the diagnostic classifications of traumatic dental injuries. Dent Traumatol. 2006 Apr;22(2):71-6. doi: 10.1111/j.1600-9657.2006.00342.x. PMID 16499629
- [Background] Hermann NV, Lauridsen E, Ahrensburg SS, Gerds TA, Andreasen JO. Periodontal healing complications following extrusive and lateral luxation in the permanent dentition: a longitudinal cohort study. Dent Traumatol. 2012 Oct;28(5):394-402. doi: 10.1111/edt.12000. Epub 2012 Sep 12. PMID 22971023
- [Background] Spinas E, Pipi L, Dettori C. Extrusive Luxation Injuries in Young Patients: A Retrospective Study with 5-Year Follow-Up. Dent J (Basel). 2020 Dec 16;8(4):136. doi: 10.3390/dj8040136. PMID 33339132
- [Background] Nikoui M, Kenny DJ, Barrett EJ. Clinical outcomes for permanent incisor luxations in a pediatric population. III. Lateral luxations. Dent Traumatol. 2003 Oct;19(5):280-5. doi: 10.1034/j.1600-9657.2003.00209.x. PMID 14708653
- [Background] Ferrazzini Pozzi EC, von Arx T. Pulp and periodontal healing of laterally luxated permanent teeth: results after 4 years. Dent Traumatol. 2008 Dec;24(6):658-62. doi: 10.1111/j.1600-9657.2008.00687.x. PMID 19021659
- [Background] Flores MT, Andersson L, Andreasen JO, Bakland LK, Malmgren B, Barnett F, Bourguignon C, DiAngelis A, Hicks L, Sigurdsson A, Trope M, Tsukiboshi M, von Arx T; International Association of Dental Traumatology. Guidelines for the management of traumatic dental injuries. I. Fractures and luxations of permanent teeth. Dent Traumatol. 2007 Apr;23(2):66-71. doi: 10.1111/j.1600-9657.2007.00592.x. PMID 17367451
- [Background] Gungor HC, Cengiz SB, Altay N. Immediate surgical repositioning following intrusive luxation: a case report and review of the literature. Dent Traumatol. 2006 Dec;22(6):340-4. doi: 10.1111/j.1600-9657.2005.00356.x. PMID 17073929
- [Background] Strobl H, Haas M, Norer B, Gerhard S, Emshoff R. Evaluation of pulpal blood flow after tooth splinting of luxated permanent maxillary incisors. Dent Traumatol. 2004 Feb;20(1):36-41. doi: 10.1046/j.1600-4469.2003.00223.x. PMID 14998413
- [Background] Emshoff R, Emshoff I, Moschen I, Strobl H. Diagnostic characteristics of pulpal blood flow levels associated with adverse outcomes of luxated permanent maxillary incisors. Dent Traumatol. 2004 Oct;20(5):270-5. doi: 10.1111/j.1600-9657.2004.00281.x. PMID 15355386
- [Background] Spinas E, Pipi L, Mezzena S, Giannetti L. Use of Orthodontic Methods in the Treatment of Dental Luxations: A Scoping Review. Dent J (Basel). 2021 Feb 4;9(2):18. doi: 10.3390/dj9020018. PMID 33557060
- [Background] Soriano EP, Caldas Ade F Jr, Diniz De Carvalho MV, Amorim Filho Hde A. Prevalence and risk factors related to traumatic dental injuries in Brazilian schoolchildren. Dent Traumatol. 2007 Aug;23(4):232-40. doi: 10.1111/j.1600-9657.2005.00426.x. PMID 17635357
- [Background] Martins VM, Sousa RV, Rocha ES, Leite RB, Paiva SM, Granville-Garcia AF. Dental trauma among Brazilian schoolchildren: prevalence, treatment and associated factors. Eur Arch Paediatr Dent. 2012 Oct;13(5):232-7. doi: 10.1007/BF03262876. PMID 23043878
- [Background] Hamdan MA, Rajab LD. Traumatic injuries to permanent anterior teeth among 12-year-old schoolchildren in Jordan. Community Dent Health. 2003 Jun;20(2):89-93. PMID 12828268
- [Background] Soriano EP, Caldas Ade F Jr, De Carvalho MV, Caldas KU. Relationship between traumatic dental injuries and obesity in Brazilian schoolchildren. Dent Traumatol. 2009 Oct;25(5):506-9. doi: 10.1111/j.1600-9657.2009.00828.x. PMID 19754696
- [Background] Navabazam A, Farahani SS. Prevalence of traumatic injuries to maxillary permanent teeth in 9- to 14-year-old school children in Yazd, Iran. Dent Traumatol. 2010 Apr;26(2):154-7. doi: 10.1111/j.1600-9657.2009.00861.x. Epub 2010 Jan 19. PMID 20089070
- [Background] Borssen E, Holm AK. Treatment of traumatic dental injuries in a cohort of 16-year-olds in northern Sweden. Endod Dent Traumatol. 2000 Dec;16(6):276-81. doi: 10.1034/j.1600-9657.2000.016006276.x. PMID 11202894
- [Background] von Arx T, Filippi A, Buser D. Splinting of traumatized teeth with a new device: TTS (Titanium Trauma Splint). Dent Traumatol. 2001 Aug;17(4):180-4. doi: 10.1034/j.1600-9657.2001.170408.x. PMID 11585145
- [Background] Petersson EE, Andersson L, Sorensen S. Traumatic oral vs non-oral injuries. Swed Dent J. 1997;21(1-2):55-68. PMID 9178450
- [Background] Andersson L. Epidemiology of traumatic dental injuries. Pediatr Dent. 2013 Mar-Apr;35(2):102-5. PMID 23635975
- [Background] Gabris K, Tarjan I, Rozsa N. Dental trauma in children presenting for treatment at the Department of Dentistry for Children and Orthodontics, Budapest, 1985-1999. Dent Traumatol. 2001 Jun;17(3):103-8. doi: 10.1034/j.1600-9657.2001.017003103.x. PMID 11499758
- [Background] Zerman N, Cavalleri G. Traumatic injuries to permanent incisors. Endod Dent Traumatol. 1993 Apr;9(2):61-4. doi: 10.1111/j.1600-9657.1993.tb00661.x. PMID 8404697
- [Background] Fakhruddin KS, Lawrence HP, Kenny DJ, Locker D. Etiology and environment of dental injuries in 12- to 14-year-old Ontario schoolchildren. Dent Traumatol. 2008 Jun;24(3):305-8. doi: 10.1111/j.1600-9657.2007.00548.x. Epub 2008 Apr 9. PMID 18410389
- [Background] Petti S, Glendor U, Andersson L. World traumatic dental injury prevalence and incidence, a meta-analysis-One billion living people have had traumatic dental injuries. Dent Traumatol. 2018 Apr;34(2):71-86. doi: 10.1111/edt.12389. PMID 29455471
- [Background] Tewari N, Mathur VP, Siddiqui I, Morankar R, Verma AR, Pandey RM. Prevalence of traumatic dental injuries in India: A systematic review and meta-analysis. Indian J Dent Res. 2020 Jul-Aug;31(4):601-614. doi: 10.4103/ijdr.IJDR_953_19. PMID 33107464
- [Background] Berthold C, Holst S, Schmitt J, Goellner M, Petschelt A. An evaluation of the Periotest method as a tool for monitoring tooth mobility in dental traumatology. Dent Traumatol. 2010 Apr;26(2):120-8. doi: 10.1111/j.1600-9657.2009.00860.x. Epub 2010 Jan 11. PMID 20070346
- [Background] Levander E, Malmgren O. Long-term follow-up of maxillary incisors with severe apical root resorption. Eur J Orthod. 2000 Feb;22(1):85-92. doi: 10.1093/ejo/22.1.85. PMID 10721249
- [Background] Chakrapani S, Goutham M, Krishnamohan T, Anuparthy S, Tadiboina N, Rambha S. Periotest values: Its reproducibility, accuracy, and variability with hormonal influence. Contemp Clin Dent. 2015 Jan-Mar;6(1):12-5. doi: 10.4103/0976-237X.149284. PMID 25684904
- [Background] Laster L, Laudenbach KW, Stoller NH. An evaluation of clinical tooth mobility measurements. J Periodontol. 1975 Oct;46(10):603-7. doi: 10.1902/jop.1975.46.10.603. PMID 1058939
- [Background] Schulte W, d'Hoedt B, Lukas D, Maunz M, Steppeler M. Periotest for measuring periodontal characteristics--correlation with periodontal bone loss. J Periodontal Res. 1992 May;27(3):184-90. doi: 10.1111/j.1600-0765.1992.tb01667.x. PMID 1608031
- [Background] Berthold C, Auer FJ, Potapov S, Petschelt A. Influence of wire extension and type on splint rigidity--evaluation by a dynamic and a static measuring method. Dent Traumatol. 2011 Dec;27(6):422-31. doi: 10.1111/j.1600-9657.2011.01033.x. Epub 2011 Jul 26. PMID 21790987
- [Background] Kwan SC, Johnson JD, Cohenca N. The effect of splint material and thickness on tooth mobility after extraction and replantation using a human cadaveric model. Dent Traumatol. 2012 Aug;28(4):277-81. doi: 10.1111/j.1600-9657.2011.01086.x. Epub 2011 Nov 23. PMID 22107132
- [Background] Oikarinen K, Andreasen JO, Andreasen FM. Rigidity of various fixation methods used as dental splints. Endod Dent Traumatol. 1992 Jun;8(3):113-9. doi: 10.1111/j.1600-9657.1992.tb00447.x. PMID 1289069
- [Background] Berthold C, Auer FJ, Potapov S, Petschelt A. In vitro splint rigidity evaluation--comparison of a dynamic and a static measuring method. Dent Traumatol. 2011 Dec;27(6):414-21. doi: 10.1111/j.1600-9657.2011.01034.x. Epub 2011 Jul 26. PMID 21790988
- [Background] Azami-Aghdash S, Ebadifard Azar F, Pournaghi Azar F, Rezapour A, Moradi-Joo M, Moosavi A, Ghertasi Oskouei S. Prevalence, etiology, and types of dental trauma in children and adolescents: systematic review and meta-analysis. Med J Islam Repub Iran. 2015 Jul 10;29(4):234. eCollection 2015. PMID 26793672
- [Background] Lam R. Epidemiology and outcomes of traumatic dental injuries: a review of the literature. Aust Dent J. 2016 Mar;61 Suppl 1:4-20. doi: 10.1111/adj.12395. PMID 26923445
- [Background] Schatz JP, Hakeberg M, Ostini E, Kiliaridis S. Prevalence of traumatic injuries to permanent dentition and its association with overjet in a Swiss child population. Dent Traumatol. 2013 Apr;29(2):110-4. doi: 10.1111/j.1600-9657.2012.01150.x. Epub 2012 May 24. PMID 22624850
- [Background] Magno MB, Neves AB, Ferreira DM, Pithon MM, Maia LC. The relationship of previous dental trauma with new cases of dental trauma. A systematic review and meta-analysis. Dent Traumatol. 2019 Feb;35(1):3-14. doi: 10.1111/edt.12449. Epub 2018 Nov 5. PMID 30307124
- [Background] Lin S, Emodi O, Abu El-Naaj I. Splinting of an injured tooth as part of emergency treatment. Dent Traumatol. 2008 Jun;24(3):370-2. doi: 10.1111/j.1600-9657.2007.00530.x. PMID 18489488
- [Background] Silva RAB, Vieira HAO, de Gregorio C, Cohenca N, Lucisano MP, Pucinelli CM, Paula-Silva FWG, Nelson-Filho P, Romano FL, Assed Bezerra Silva L. Periodontal ligament repair after active splinting of replanted dogs' teeth. Dent Traumatol. 2021 Dec;37(6):758-771. doi: 10.1111/edt.12698. Epub 2021 Jul 1. PMID 34198370
- [Background] Ramos-Jorge ML, Ramos-Jorge J, Mota-Veloso I, Oliva KJ, Zarzar PM, Marques LS. Parents' recognition of dental trauma in their children. Dent Traumatol. 2013 Aug;29(4):266-71. doi: 10.1111/edt.12005. Epub 2012 Oct 16. PMID 23067276
- [Background] Andreasen JO, Lauridsen E, Gerds TA, Ahrensburg SS. Dental Trauma Guide: a source of evidence-based treatment guidelines for dental trauma. Dent Traumatol. 2012 Apr;28(2):142-7. doi: 10.1111/j.1600-9657.2011.01059.x. Epub 2012 Jan 25. PMID 22272918
- [Background] Burcak Cengiz S, Stephan Atac A, Cehreli ZC. Biomechanical effects of splint types on traumatized tooth: a photoelastic stress analysis. Dent Traumatol. 2006 Jun;22(3):133-8. doi: 10.1111/j.1600-9657.2006.00339.x. PMID 16643288
- [Background] Heithersay GS. Life cycles of traumatized teeth: long-term observations from a cohort of dental trauma victims. Aust Dent J. 2016 Mar;61 Suppl 1:120-7. doi: 10.1111/adj.12403. PMID 26923453
- [Background] Andreasen JO, Andreasen FM, Skeie A, Hjorting-Hansen E, Schwartz O. Effect of treatment delay upon pulp and periodontal healing of traumatic dental injuries -- a review article. Dent Traumatol. 2002 Jun;18(3):116-28. doi: 10.1034/j.1600-9657.2002.00079.x. PMID 12110104
- [Background] Pelka M, Berthold C, van Waes H. Late reposition of a lateral luxated maxillary incisor with an immature apex. Dent Traumatol. 2009 Oct;25(5):550-4. doi: 10.1111/j.1600-9657.2009.00814.x. PMID 19754701
- [Background] Lauridsen E, Hermann NV, Gerds TA, Ahrensburg SS, Kreiborg S, Andreasen JO. Combination injuries 3. The risk of pulp necrosis in permanent teeth with extrusion or lateral luxation and concomitant crown fractures without pulp exposure. Dent Traumatol. 2012 Oct;28(5):379-85. doi: 10.1111/j.1600-9657.2011.01100.x. Epub 2012 Jan 11. PMID 22233180
- [Background] Berthold C, Auer FJ, Potapov S, Petschelt A. Development of new artificial models for splint rigidity evaluation. Dent Traumatol. 2011 Oct;27(5):356-67. doi: 10.1111/j.1600-9657.2011.01010.x. Epub 2011 May 27. PMID 21615861
- [Background] Mazzoleni S, Meschia G, Cortesi R, Bressan E, Tomasi C, Ferro R, Stellini E. In vitro comparison of the flexibility of different splint systems used in dental traumatology. Dent Traumatol. 2010 Feb;26(1):30-6. doi: 10.1111/j.1600-9657.2009.00843.x. PMID 20089059
- [Background] Oikarinen K. Functional fixation for traumatically luxated teeth. Endod Dent Traumatol. 1987 Oct;3(5):224-8. doi: 10.1111/j.1600-9657.1987.tb00627.x. No abstract available. PMID 3479321
- [Background] Baena Lopes M, Romero Felizardo K, Danil Guiraldo R, Fancio Sella K, Ramos Junior S, Gonini Junior A, Bittencourt Berger S. Photoelastic stress analysis of different types of anterior teeth splints. Dent Traumatol. 2021 Apr;37(2):256-263. doi: 10.1111/edt.12618. Epub 2020 Dec 12. PMID 33180992
- [Background] Vilela ABF, Soares PBF, Beaini TL, Versluis A, Soares CJ. Splint stiffness and extension effects on a simulated avulsed permanent incisor-A patient-specific finite element analysis. Dent Traumatol. 2022 Feb;38(1):53-61. doi: 10.1111/edt.12705. Epub 2021 Jul 26. PMID 34309197
- [Background] Bauss O, Schwestka-Polly R, Schilke R, Kiliaridis S. Effect of different splinting methods and fixation periods on root development of autotransplanted immature third molars. J Oral Maxillofac Surg. 2005 Mar;63(3):304-10. doi: 10.1016/j.joms.2004.06.056. PMID 15742278
- [Background] Cehreli ZC, Lakshmipathy M, Yazici R. Effect of different splint removal techniques on the surface roughness of human enamel: a three-dimensional optical profilometry analysis. Dent Traumatol. 2008 Apr;24(2):177-82. doi: 10.1111/j.1600-9657.2007.00491.x. PMID 18352920
- [Background] Dettwiler C, Meller C, Eggmann F, Saccardin F, Kuhl S, Filippi A, Krastl G, Weiger R, Connert T. Evaluation of a Fluorescence-aided Identification Technique (FIT) for removal of composite bonded trauma splints. Dent Traumatol. 2018 Oct;34(5):353-359. doi: 10.1111/edt.12425. Epub 2018 Aug 24. PMID 29983006
- [Background] Franz F, Potapov S, Petschelt A, Berthold C. Influence of adhesive point dimension and splint type on splint rigidity--evaluation by the dynamic Periotest method. Dent Traumatol. 2013 Jun;29(3):203-11. doi: 10.1111/j.1600-9657.2012.01164.x. Epub 2012 Jul 22. PMID 22816496
- [Background] Kahler B, Heithersay GS. An evidence-based appraisal of splinting luxated, avulsed and root-fractured teeth. Dent Traumatol. 2008 Feb;24(1):2-10. doi: 10.1111/j.1600-9657.2006.00480.x. PMID 18173657
- [Background] Oikarinen K. Tooth splinting: a review of the literature and consideration of the versatility of a wire-composite splint. Endod Dent Traumatol. 1990 Dec;6(6):237-50. doi: 10.1111/j.1600-9657.1990.tb00426.x. PMID 2094598
- [Background] de Souza FI, Poi WR, da Silva VF, Martini AP, Melo RA, Panzarini SR, Rocha EP. Stress distribution in delayed replanted teeth splinted with different orthodontic wires: a three-dimensional finite element analysis. Dent Traumatol. 2015 Jun;31(3):190-5. doi: 10.1111/edt.12159. Epub 2015 Jan 21. PMID 25604805
- [Background] Kahler B, Hu JY, Marriot-Smith CS, Heithersay GS. Splinting of teeth following trauma: a review and a new splinting recommendation. Aust Dent J. 2016 Mar;61 Suppl 1:59-73. doi: 10.1111/adj.12398. PMID 26923448
- [Background] Filippi A, von Arx T, Lussi A. Comfort and discomfort of dental trauma splints - a comparison of a new device (TTS) with three commonly used splinting techniques. Dent Traumatol. 2002 Oct;18(5):275-80. doi: 10.1034/j.1600-9657.2002.00121.x. PMID 12427202
- [Background] Ben Hassan MW, Andersson L, Lucas PW. Stiffness characteristics of splints for fixation of traumatized teeth. Dent Traumatol. 2016 Apr;32(2):140-5. doi: 10.1111/edt.12234. Epub 2015 Oct 8. PMID 26449180
- [Background] von Arx T. Splinting of traumatized teeth with focus on adhesive techniques. J Calif Dent Assoc. 2005 May;33(5):409-14. PMID 16033040
- [Background] Berthold C, Thaler A, Petschelt A. Rigidity of commonly used dental trauma splints. Dent Traumatol. 2009 Jun;25(3):248-55. doi: 10.1111/j.1600-9657.2008.00683.x. PMID 19583572
- [Background] von Arx T, Filippi A, Lussi A. Comparison of a new dental trauma splint device (TTS) with three commonly used splinting techniques. Dent Traumatol. 2001 Dec;17(6):266-74. doi: 10.1034/j.1600-9657.2001.170605.x. PMID 11766094
- [Background] Ramesh P, Mathew S, Murthy SB, George JV, Hegde S, Premkumar R. Efficacy of Ribbond and a fibre post on the fracture resistance of reattached maxillary central incisors with two fracture patterns: a comparative in vitro study. Dent Traumatol. 2016 Apr;32(2):110-5. doi: 10.1111/edt.12223. Epub 2015 Sep 10. PMID 26361080
- [Background] Yildirim Oz G, Ataoglu H, Kir N, Karaman AI. An alternative method for splinting of traumatized teeth: case reports. Dent Traumatol. 2006 Dec;22(6):345-9. doi: 10.1111/j.1600-9657.2005.00364.x. PMID 17073930
- [Background] Friskopp J, Blomlof L, Soder PO. Fiber glass splints. J Periodontol. 1979 Apr;50(4):193-6. doi: 10.1902/jop.1979.50.4.193. PMID 286040
- [Background] Qin M, Ge L, Bai R. Use of a removable splint in the treatment of subluxated, luxated and root fractured anterior permanent teeth in children. Dent Traumatol. 2002 Apr;18(2):81-5. doi: 10.1034/j.1600-9657.2002.180207.x. PMID 12184217
- [Background] Traebert J, Bittencourt DD, Peres KG, Peres MA, de Lacerda JT, Marcenes W. Aetiology and rates of treatment of traumatic dental injuries among 12-year-old school children in a town in southern Brazil. Dent Traumatol. 2006 Aug;22(4):173-8. doi: 10.1111/j.1600-9657.2006.00359.x. PMID 16872385
- [Background] Ebeleseder KA, Glockner K, Pertl C, Stadtler P. Splints made of wire and composite: an investigation of lateral tooth mobility in vivo. Endod Dent Traumatol. 1995 Dec;11(6):288-93. doi: 10.1111/j.1600-9657.1995.tb00506.x. PMID 8617165
- [Background] Negri MR, Panzarini SR, Poi WR, Sonoda CK, Manfrin TM, Vendrame dos Santos CL. Use of a cyanoacrylate ester adhesive for splinting of replanted teeth. Dent Traumatol. 2008 Dec;24(6):695-7. doi: 10.1111/j.1600-9657.2008.00629.x. PMID 19021667
- [Background] Lee JY, Divaris K. Hidden consequences of dental trauma: the social and psychological effects. Pediatr Dent. 2009 Mar-Apr;31(2):96-101. PMID 19455926
- [Background] Sonnenschein SK, Ziegler P, Ciardo A, Ruetters M, Krisam J, Kim TS. The impact of splinting mobile mandibular incisors on Oral Health-Related Quality of Life-Preliminary observations from a randomized clinical trial. J Clin Periodontol. 2021 Jun;48(6):816-825. doi: 10.1111/jcpe.13454. Epub 2021 Mar 17. PMID 33751644